CLINICAL TRIAL: NCT00980863
Title: Effects of a Lifestyle Intervention on Body Mass Index in Patients With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Waldemar Greil, Privatklinik Sanatorium Kilchberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LQ-bip
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle intervention to increase physical activity (Active Comparator)
  Interventions: Behavioral: lifestyle intervention to increase physical activity
- waiting control group (No Intervention)
  Interventions: Behavioral: lifestyle intervention to increase physical activity

INTERVENTIONS:
Behavioral: lifestyle intervention to increase physical activity

SUMMARY:
Patients with bipolar disorder are at increased risk of weight gain, which in turn, increases the risk for somatic disease and non-adherence to maintenance therapy. Therefore, interventions addressing weight gain are expedient for the management of this disorder. The investigators set out to evaluate the effects of a lifestyle intervention on body mass index, cardiovascular, glycemic and metabolic parameters in patients with bipolar disorder under mood stabilizing pharmacological treatment. 50 outpatients with bipolar disorder under mood stabilizing treatment participated in a randomized controlled trial (waiting control group N=24 and multimodal lifestyle intervention N=26). Each experimental group consisted of two cohorts. The intervention lasted five months and consisted of eleven group sessions and weekly fitness training. Body Mass Index (BMI), body weight as well as cardiovascular, glycemic and metabolic parameters were determined as baseline (March and September 2005) and after five (July 2005 and January 2006) and eleven months (January and July 2006).

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 70 years of age were considered for inclusion if they:

  1. fulfilled the diagnostic criteria for bipolar disorder according to DSM-IV-TR,27;
  2. were on treatment with medication for at least three months with one of the following substances: lithium, valproic acid carbamazepine, oxcarbazepine, olanzapine, quetiapine, risperidone, amisulpride; and
  3. were not underweight (BMI > 20 kg/m2).

Exclusion Criteria:

* Pregnancy
* Actual breast feeding
* A diagnosis of anorexia nervosa or bulimia nervosa
* Diabetes type I or II or another serious physical disease
* Use of substances that reduce weight (e.g., topiramate, lamotrigine as mood stabilizer in monotherapy)
* Participants with comorbidity of acute psychosis, drug addiction, personality disorder, suicidal tendencies or a current severe manic or depressive episode were excluded only if attending the program was not possible due to the respective disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
BMI | 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar Greil, Professor, Principal Investigator — Sanatorium Kilchberg, Switzerland
Locations (1):
- Sanatorium Kilchberg, Zurich, Switzerland

REFERENCES:
- [Derived] Gillhoff K, Gaab J, Emini L, Maroni C, Tholuck J, Greil W. Effects of a multimodal lifestyle intervention on body mass index in patients with bipolar disorder: a randomized controlled trial. Prim Care Companion J Clin Psychiatry. 2010;12(5):PCC.09m00906. doi: 10.4088/PCC.09m00906yel. PMID 21274359